CLINICAL TRIAL: NCT07401914
Title: The Effect of Anesthesia Protocols Used in Gastrointestinal Endoscopy Procedures in Adolescents on the Outcome
Brief Title: Ketodex Versus Ketofol in Adolescent Gastrointestinal Endoscopy
Status: Not yet recruiting | Type: Observational
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Dilek Yeniay, Anesthesiology and Reanimation physician, Giresun University
Other Study IDs: GOKAEK 2025/13/19
Record Dates: First submitted 2026-01-27; First posted 2026-02-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Procedural Sedation; Gastrointestinal Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group D (Ketodex): Patients receiving ketamine-dexmedetomidine sedation according to routine clinical practice.
  Interventions: Drug: Ketodex
- Group P (Ketofol): Patients receiving ketamine-propofol sedation according to routine clinical practice.
  Interventions: Drug: Ketofol

INTERVENTIONS:
Drug: Ketodex — Administered as part of standard institutional anesthesia practice.
  Other Names: Ketamine-Dexmedetomidine
  Groups: Group D (Ketodex)
Drug: Ketofol — Administered as part of standard institutional anesthesia practice.
  Other Names: Ketamine-Propofol
  Groups: Group P (Ketofol)

SUMMARY:
Gastrointestinal endoscopic procedures in adolescents require effective sedoanalgesia to ensure procedural comfort and prevent agitation. Pain control is an essential component of these procedures, and current practice commonly involves low-dose combinations of anesthetic agents. Sedoanalgesia protocols are selected according to patient characteristics and the anesthesiologist's clinical experience. This prospective observational study aims to compare the effects of ketodex and ketofol on intraoperative procedural comfort, postoperative recovery, and patient satisfaction in adolescents undergoing gastrointestinal endoscopy.

DETAILED DESCRIPTION:
Gastrointestinal endoscopic (GE) procedures require the use of sedoanalgesic agents to ensure patient comfort and procedural safety. In adolescent patients, deep sedation is often necessary to provide adequate procedural comfort and to prevent agitation. Additionally, GE procedures are inherently painful and require the use of analgesic medications as part of routine practice. The scientifically accepted approach involves the use of low-dose combinations of different anesthetic agents. The selection of the sedoanalgesia protocol during the procedure is shaped by patient characteristics as well as the experience and preference of the attending anesthesiologist.

The aim of this study is to evaluate the effects of routinely used sedoanalgesia protocols, specifically ketodex and ketofol, on intraoperative procedural comfort, postoperative recovery, and patient satisfaction in adolescent patients undergoing gastrointestinal endoscopy.

ELIGIBILITY:
Inclusion Criteria:

ASA I-II, adolescents aged 10-18 years undergoing elective gastrointestinal endoscopic procedures

Exclusion Criteria:

* Emergency cases
* Children under 10 years of age
* Children with mental retardation
* Children whose parents refuse to participate in the study and children who do not consent to participate themselves
* Children with known allergy, hypersensitivity, intolerance or contraindication to any of the sedoanalgesic drugs used

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescent patients scheduled to undergo gastrointestinal endoscopic procedures under sedation as part of routine clinical care will be included in the study. Patients will receive either ketamine-dexmedetomidine (ketodex) or ketamine-propofol (ketofol) sedation according to standard institutional practice and the preference of the attending anesthesiologist.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative patient comfort assessed by Ramsey Sedation Scale | During the intraoperative period
  Intraoperative patient comfort was evaluated using the Ramsey Sedation Scale, a 6-point clinical scale assessing the level of sedation and patient responsiveness.
  The scale ranges from 1 to 6, where lower scores indicate agitation or anxiety and higher scores indicate deeper sedation and better patient comfort.
Intraoperative additional anesthetic drug requirement | During the intraoperative period
  The requirement for additional anesthetic medication administered during the intraoperative period was recorded.
  Additional anesthetic use was determined based on clinical signs of inadequate sedation or patient discomfort as judged by the attending anesthesiologist.

SECONDARY OUTCOMES:
Postoperative recovery time assessed by recovery score | From the end of surgery until discharge from the postanesthesia care unit, assessed up to 24 hours postoperatively.
  Postoperative recovery time was assessed using a standardized recovery score evaluating the patient's level of consciousness and readiness for discharge from the postanesthesia care unit.
  Higher scores indicate better recovery status.
Emergence agitation assessed by emergence agitation score | From the end of anesthesia until discharge from the postanesthesia care unit, assessed up to 24 hours postoperatively.
  Emergence agitation was evaluated using a validated emergence agitation scoring system.
  The scale assesses the severity of agitation during emergence from anesthesia, with higher scores indicating greater levels of agitation.between the ketodex and ketofol groups during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Dilek YENİAY, Principal Investigator — Department of Anesthesiolgy, Giresun University

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and confidentiality considerations.